CLINICAL TRIAL: NCT05640635
Title: Inflammation During ECMO Therapy and ECMO Weaning
Acronym: ECMOWean
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECMOWean
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Extracorporal membrane oxygenation; Extracorporal membrane oxygenation weaning; Ventilation therapy
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilator weaning first (Active Comparator)
  Interventions: Procedure: Ventilator weaning first
- ECMO weaning first (Active Comparator)
  Interventions: Procedure: ECMO weaning first

INTERVENTIONS:
Procedure: Ventilator weaning first — Ventilator weaning initiated and completed before start of ECMO weaning.
  Arms: Ventilator weaning first
Procedure: ECMO weaning first — ECMO weaning initiated and completed before start of ventilator weaning.
  Arms: ECMO weaning first

SUMMARY:
The goal of this interventional clinical trial is to compare patients who undergo ECMO therapy for treatment of acute respiratory distress syndrome (ARDS) and a randomized into one of two possible weaning strategy groups.

Group 1: Weaning from ventilator occurs before ECMO weaning.

Group 2: Weaning from ECMO occurs before weaning from ventilator.

This study investigates which one of these strategies is more indulgent for the lung, and leads to less inflammation and therefore less potential side effects and an overall more favourable clinical course.

As a primary criterion, measure of IL-6 in blood samples will beused. As secondary criterions, SOFA score at various time points, ventilation pressures, lung injury score (LIS), length of stay in the intensive care unit, and ventilator-associated pneumonia as well as levels of inflammatory cells and cytokines in both blood samples and bronchoalveolar lavage at different time points will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory distress syndrome (ARDS) according to the Berlin Definition (PaO2/FiO2 < 100) and treatment with veno-venous ECMO (vvECMO)
* Hemodynamic stability
* Lung compliance did not change/improved during the last 24 hours
* Tidal volume did not change/improved during the last 24 hours with a PEEP of 10 cmH20 or above
* Consent of the patient or their legal representative

Exclusion Criteria:

* Age < 18 years
* Artificial ventilation for more than 7 days prior
* Patient, legal representative or doctors decided against an unrestricted intensive care treatment
* Positive pregnancy test at time of screening
* Cardiac failure requiring veno-arterial ECMO therapy
* Chronic respiratory insufficiency requiring long-term oxygen treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
IL-6 concentration (blood samples) | For the duration of the ICU stay, or a maximum of 60 days.
  Daily control of above mentioned parameter.

SECONDARY OUTCOMES:
SOFA-Score | For the duration of the ICU stay, or a maximum of 60 days at indicated time points as described above..
  Sequential organ failure assessement score evaluated at days 1-14, 28, and 60.
Ventilation pressures | For the duration of the artificial ventilation, or a maximum of 60 days.
  Pressures applied to the lung during artificial ventilation
Murray Lung Injury Score (LIS) | For the duration of the ICU stay, or a maximum of 60 days.
  Assessement of severity of lung damage by the established Lung Injury Score by Murray (Min Value is 0, healthy and Max Value is 20, severly diseased)
Length of stay in the intensive care unit | For the duration of the ICU stay, or a maximum of 60 days.
  Length of stay in the intensive care unit.
Ventilator-associated pneumonia | For the duration of the ICU stay, or a maximum of 60 days.
  Occurence/incidence of ventilator-associated pneumonia.
Cytokines and inflammatory cells in blood samples (IL-1beta, Il-10 and TNF-alpha) | For the duration of the ICU stay, or a maximum of 60 days.
  Collection of blood samples at various times points for further analysis.
Cytokines and inflammatory cells in bronchoalveolar lavage (IL-1beta, Il-10 and TNF-alpha) | For the duration of the ICU stay, or a maximum of 60 days.
  Collection of bronchoalveolar lavage samples at various times points for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, Prof., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany